CLINICAL TRIAL: NCT01198795
Title: An Open-label Long-term Study of Escitalopram in Children 7 to 11 Years of Age With Major Depressive Disorder
Brief Title: Safety Study of Escitalopram in Children 7 to 11 Years of Age With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT-MD-55
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-01

CONDITIONS: Major Depressive Disorder
Keywords: depression; major depressive disorder; escitalopram; Lexapro; pediatric
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Flexible-dose 10mg-20mg once-daily oral (10mg tablets) dose of escitalopram
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Patients who meet eligibility criteria will receive open-label escitalopram. 10-20mg oral administration (10mg tablets) once daily for 24-weeks with a 2-week downtaper period.
  Other Names: Lexapro

SUMMARY:
This study will evaluate the long-term safety and tolerability of escitalopram (Lexapro) in children 7 to 11 years of age with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 7 to 11 years of age, inclusive
* Current diagnosis of MDD based on DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision) criteria as confirmed by K-SADS-PL (Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime) with a minimum duration of 6 weeks
* Patient's parent(s), guardian(s), or LAR(s) is capable of providing information about his or her condition, provides informed consent, and agrees to accompany the patient to all study visits. (Preferably the same parent, guardian, or LAR will accompany the patient to all study visits)
* Patient's family is sufficiently organized and stable to guarantee adequate safety monitoring

Exclusion Criteria:

* Current principal DSM-IV-TR-based diagnosis of an axis I disorder other than MDD that was the primary focus of treatment
* Patients with a diagnosis of conduct disorder will not be allowed to participate in this study
* Current diagnosis of mental retardation, dementia, or amnestic or other cognitive disorders based on DSM-IV-TR criteria
* History of allergy, intolerance, or hypersensitivity to escitalopram, citalopram, or other drugs of the same class
* Imminent risk of injuring self or others or causing significant damage to property, as judged by the PI
* Suicide risk as determined by meeting any of the following criteria:

  * Any suicide attempt
  * Significant risk, as judged by the PI, based on the psychiatric interview or information collected in the Columbia-Suicide Severity Rating Scale (C-SSRS)

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suneeta Ahuja, PhD, Study Chair — Forest Laboratories
Locations (16):
- United States (16):
  - Forest Investigative Site 001, Dothan, Alabama
  - Forest Investigative Site 006, San Diego, California
  - Forest Investigative Site 018, Santa Ana, California
  - Forest Investigative Site 008, Washington D.C., District of Columbia
  - Forest Investigative Site 013, Jacksonville Beach, Florida
  - Forest Investigative Site 017, Atlanta, Georgia
  - Forest Investigative Site 004, Overland Park, Kansas
  - Forest Investigative Site 011, Creve Coeur, Missouri
  - Forest Investigative Site 007, Omaha, Nebraska
  - Forest Investigative Site 002, Cleveland, Ohio
  - Forest Investigative Site 012, Oklahoma City, Oklahoma
  - Forest Investigative Site 003, Philadelphia, Pennsylvania
  - Forest Investigative Site 010, Dallas, Texas
  - Forest Investigative Site 014, Clinton, Utah
  - Forest Investigative Site 005, Bellevue, Washington
  - Forest Investigative Site 015, Kirkland, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred at 16 studies sites located in the US from October of 2010 to August of 2012.
Pre-assignment Details: All patients completed a 1-week no-drug screening period before beginning treatment with study drug.
Groups:
- Escitalopram: Flexible-dose 10mg-20mg once-daily oral (10mg tablets) dose of escitalopram for 24-weeks, with a 2-week downtaper period.
Period: Overall Study
Arm/Group | Escitalopram
Started | 162
Completed | 80
Not Completed | 82
Not completed — Did not meet InclusionExclusion criteria | 30
Not completed — Withdrawal by Subject | 17
Not completed — Lost to Follow-up | 15
Not completed — Adverse Event | 9
Not completed — Lack of Efficacy | 5
Not completed — Protocol Violation | 2
Not completed — Other Reason | 4

BASELINE CHARACTERISTICS:
Population: A total of 162 unique patients were enrolled in the study. Of these, 118 patients received at least 1 dose of investigational product to comprise the Safety Population. All 118 patients in the Safety Population also had at least 1 postbaseline efficacy assessment, and comprise the Intent To Treat (ITT) Population.
Arm/Group | Escitalopram
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.4 (1.2)
Age, Customized [Number; unit: participants]
  Ages 7 Years to 8 Years | 31
  Ages 9 Years to 10 Years | 62
  Age 11 Years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 65
Race/Ethnicity, Customized [Number; unit: participants]
  White | 85
  Black | 26
  Asian | 1
  American Indian or Alaska Native | 1
  Native Hawaiian or Other Pacific Islander | 1
  Other | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 102
Region of Enrollment [Number; unit: participants]
  United States | 118
Weight, mean [Mean (Standard Deviation); unit: kg] | 42.71 (16.67)
Height, mean [Mean (Standard Deviation); unit: cm] | 141.27 (10.22)
BMI(Body Mass Index), mean [Mean (Standard Deviation); unit: kg/m2] | 20.86 (5.83)

OUTCOME MEASURES:

1. Primary Outcome: Patients With Any Treatment Emergent Adverse Events (TEAEs)
Description: The number of patients who experienced one or more TEAE during the 24-week open-label treatment period or the 2-week down-taper period,
Time Frame: From Baseline (Week 0) to Week 26
Measure: Number; unit: participants
Arm/Group | Escitalopram
Number analyzed (Participants) | 118
participants | 89

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during a 28 month period from October 2010 to February 2013.
Arm/Group | Escitalopram
Serious Adverse Events (participants affected / at risk) | 2/118
Other Adverse Events (participants affected / at risk) | 59/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=118)
Mania (Psychiatric disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Escitalopram (N=118)
Abdominal pain upper (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 9
Nausea (General disorders) | 6
Vomiting (General disorders) | 7
Nasopharyngitis (Infections and infestations) | 9
Increased appetite (Metabolism and nutrition disorders) | 7
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 20
Insomnia (Psychiatric disorders) | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.